CLINICAL TRIAL: NCT06014476
Title: Psychological Symptoms and Burden in Caregivers of Patients With Disorders of Consciousness
Status: Completed | Type: Observational
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Haibo Di, Principal Investigator, Hangzhou Normal University
Other Study IDs: Hangzhou Normal University
Record Dates: First submitted 2023-08-15; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Psychological Distress; Anxiety Depression; Burden, Caregiver; Disorders of Consciousness
MeSH Terms: conditions — Caregiver Burden; Consciousness Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Caregivers of patients with disorders of consciousness, including Coma, Unresponsive Wakefulness Syndrome (UWS), and Minimally Consciousness State (MCS). And caregivers of patients emerge from the minimally conscious state (EMCS)
  Interventions: Other: questionnaires
- Control group: caregivers of patients with other disease
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Sent questionnaires to caregivers and used CRS-R to assess patients with DoC
  Other Names: Coma Recovery Scale-Revised (CRS-R)

SUMMARY:
Caregivers of patients with disorders of consciousness are highly prone to developing mental health issues. The aim of this study is to investigate the psychological symptoms and care burden of caregivers of patients with disorders of consciousness (DoC), and to examine which characteristics of patients were burden predictors to caregivers.

DETAILED DESCRIPTION:
This is a multi-center cross-sectional study in China, from August 2021 to October 2022. Patients were assessed by Coma Recovery Scale-Revised (CRS-R), and caregivers' anxiety, depression, and burden were assessed by State-Trait Anxiety Inventory Form Y (STAI), Beck Depression Inventory-II (BDI- II), and Zarit Caregiver Burden scale (ZBI). The comparison with patients' age and caregivers' age-matched subjects who were randomly selected and without DoC; intra-group comparison of caregivers for DoC was conducted. Descriptive statistics were used to illustrate the socio-demographics. One-sample t-test, independent sample t-test, one-way ANOVA, Mann-Whitney U test, and Kruskal-Wallis test were executed to detect the difference between groups due to the distribution of each variable.

ELIGIBILITY:
Inclusion Criteria:

- (1) Family caregivers without neurological, mental health, or learning disability history.

(2) Family caregiver with consciousness and capability of independently completing questionnaires.

Exclusion criteria:

1. Caregivers unwilling to participate
2. Not the dominant caregivers

Ages: 17 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Caregivers of patients with DoC and other diseases
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The prevalence of anxiety in caregivers of patients with disorders of consciousness. | Within 1 days
  We use the State-Trait Anxiety Inventory Form Y (STAI-Y) to assess the prevalence and severity degree of anxiety for caregivers of patients with disorders of consciousness (DoC)
  STAI was a self-rating scale, consisting of 40 items and divided into two subscales: 1) state anxiety (S-AI) scale includes questions 1-20, state anxiety shows the transitory unpleasant. 2) trait anxiety (T-AI) scale includes questions 21-40, trait anxiety tends to the personality trait. The cumulative score values of state anxiety and trait anxiety scales were calculated respectively, the minimum to maximum value was from 20 to 80, the higher scores mean a worse outcome.
The prevalence and severity degree of depression in caregivers of patients with disorders of consciousness. | Within 1 days
  We use the Beck Depression Inventory-II (BDI-II) to assess the prevalence and severity degree of depression for caregivers of patients with disorders of consciousness (DoC)
  BDI total score: 0-13 as no depression, 14-19 as mild depression, 20-28 as medium depression, and 29-63 as severe depression.
The prevalence and severity degree of burden in caregivers of patients with disorders of consciousness. | Within 1 days
  We use the Zarit Caregiver Burden Scale (ZBI) to assess the prevalence and severity degree of burden for caregivers of patients with disorders of consciousness (DoC)
  ZBI total score: 0-20 indicates no burden, 21-40 mild burden, 41-60 moderate burden, and 61-88 severe burden.
The predictors of anxiety in caregivers of patients with disorders of consciousness. | Within 1 days
  We choose a series of questionnaires to figure out: what are the characteristics of patients and caregivers were caregivers' anxiety predictors?
  The questionnaires include social-demographic questionnaires (including personal information of patients and caregivers e.g., age, gender, etiology, diagnosis, and so on, to record their basic information) and the State-Trait Anxiety Inventory Form Y (STAI-Y).
  We used the Independent-sample T-test, one-way ANOVA, Mann-Whitney U test, Kruskal-Wallis test, and Pearson Correlation to calculate the correlation between the characteristics of patients and caregivers and caregivers' anxiety.
The predictors of depression in caregivers of patients with disorders of consciousness. | Within 1 days
  We choose a series of questionnaires to figure out:
  (1) What are the characteristics of patients and caregivers were caregivers' depression predictors?
  The questionnaires include social-demographic questionnaires (including personal information of patients and caregivers e.g., age, gender, etiology, diagnosis, and so on, to record their basic information), and the Beck Depression Inventory-II (BDI-II).
  We used the Independent-sample T-test, one-way ANOVA, Mann-Whitney U test, Kruskal-Wallis test, and Pearson Correlation to calculate the correlation between the characteristics of patients and caregivers and caregivers' depression.
The predictors of burden in caregivers of patients with disorders of consciousness. | Within 1 days
  We choose a series of questionnaires to figure out:
  (1) What are the characteristics of patients and caregivers were caregivers' burden predictors?
  The questionnaires include social-demographic questionnaires (including personal information of patients and caregivers e.g., age, gender, etiology, diagnosis, and so on, to record their basic information), and the Zarit Caregiver Burden Scale (ZBI).
  We used the Independent-sample T-test, one-way ANOVA, Mann-Whitney U test, Kruskal-Wallis test, and Pearson Correlation to calculate the correlation between the characteristics of patients and caregivers and caregivers' burden.

SECONDARY OUTCOMES:
The diagnoses of patients with disorders of consciousness (DoC) | Within 10 days
  The DoC patients were evaluated 3-5 times Coma Recovery Scale-Revised (CRS-R) within 10 days after questionnaire distribution to determine their current state of consciousness.
The relationship between patient diagnoses and caregivers' anxiety | Within 1 days
  We compare patient diagnoses (assessed by Coma Recovery Scale-Revised (CRS-R) ) and caregivers' anxiety (assessed by the State-Trait Anxiety Inventory Form Y (STAI-Y) )
  We used the one-way ANOVA to calculate the relationship between patient diagnoses and caregivers' anxiety.
The relationship between patient diagnoses and caregivers' depression | Within 1 days
  We compare patient diagnoses (assessed by Coma Recovery Scale-Revised (CRS-R) ) and caregivers' depression (assessed by the Beck Depression Inventory-II (BDI-II) )
  We used the one-way ANOVA to calculate the relationship between patient diagnoses and caregivers' depression.
The relationship between patient diagnoses and caregivers' burden | Within 1 days
  We compare patient diagnoses (assessed by Coma Recovery Scale-Revised (CRS-R) ) and caregivers' depression (assessed by the Zarit Caregiver Burden Scale (ZBI) )
  We used the one-way ANOVA to calculate the relationship between patient diagnoses and caregivers' burden.

CONTACTS AND LOCATIONS:
Overall Officials: Hao YA Wang, Study Chair — Hangzhou Normal University
Locations (1):
- International Vegetative State and Consciousness Science Institute, Hangzhou Normal University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No